CLINICAL TRIAL: NCT06017362
Title: Ensayo Clínico Para Determinar La Eficacia Y Seguridad Del Colirio De Insulina En El Tratamiento Del Ojo Seco En Pacientes Con Hipotensores Tópicos
Brief Title: Clinical Trial to Determine the Efficacy and Safety of Insulin Eye Drops in Dry Eye in Patients with Topical Hypotensors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Barbara Burgos Blasco (Other)
Responsible Party: Sponsor-Investigator, Barbara Burgos Blasco, Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22/457-EC_M
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye; Glaucoma
MeSH Terms: conditions — Dry Eye Syndromes; Glaucoma | interventions — Insulin; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin (Experimental): Topical insulin 1UI/ml 4 times a day
  Interventions: Drug: Insulin
- Placebo (artificial tears) (Placebo Comparator): Artificial tears 4 times a day
  Interventions: Drug: Artificial tear

INTERVENTIONS:
Drug: Insulin — Topical insulin 1UI/ml 4 times a day
  Arms: Insulin
Drug: Artificial tear — Artificial tears 4 times a day
  Arms: Placebo (artificial tears)

SUMMARY:
The goal of this clinical trial is to evaluate the preliminary efficacy of the use of insulin eye drops in the control of dry eye disease in patients with topical hypotensors, compared to placebo (artificial tears).

The main question aims to answer whether glaucoma patients treated with topical hypotensors could benefit from the use of insulin eye drops for the treatment of dry eye.

Participants will be assigned to one of the two treatment arms and will be required to attend four follow-up visits (baseline, 1, 3, and 6 months).

DETAILED DESCRIPTION:
Patients will be recruited in Madrid. Patients with dry eye disease and topical glaucoma treatment will be identified through the Ophthalmology clinic. They will be directly referred to a physician who is participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide written informed consent and who are able and willing to comply with all scheduled study visits and procedures.
* Patients ≥ 18 years at the screening visit.
* Ocular hypertension or glaucoma controlled with hypotensive treatment
* Diagnosis of dry eye

Exclusion Criteria:

* Uncontrolled glaucoma with expected changes in antihypertensive treatment in the next 6 months
* Changes in topical glaucoma treatment in the last 3 months
* Severe dry eye requiring immediate treatment
* Previous eye surgery, except cataract surgery more than 12 months ago
* Laser procedures less than 6 months ago
* Other concomitant ocular pathology: scarring disease of the ocular surface, uveitis, infection in the last 90 days, trauma in the last 90 days
* Eyelid disorders
* Use of contact lenses
* Other topical treatment other than dry eye and glaucoma
* Patients with a history of allergy or hypersensitivity to the study medication or any of its excipients
* Modifications in systemic immunosuppressive treatment in the last 6 months
* History of alcohol or drug abuse
* Patients who have received an experimental drug or used an experimental medical device in the 30-day period prior to the screening visit.
* Systemic pathology (cardiopulmonary pathology, connective tissue disorders, neurological or psychiatric pathology) or situation of the patient that does not allow examination (such as mental or psychomotor retardation).
* Any other disease or condition that, at the discretion of the investigator, could constitute a risk to the participant or interfere with the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Changes in dry eye symptoms from baseline to 6 months after treatment time | From baseline to 6 months after treatment
  Dry eye symptoms will be evaluated using OSDI

SECONDARY OUTCOMES:
Change of corneal staining from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Corneal staining will be evaluated on the slit-lamp and on slit-lamp images
Change in corneal aesthesiometry from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Aesthesiometry will be evaluated using Cochet Bonnet
Change in conjunctival hyperemia from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Conjunctival hyperemia will be evaluated using Keratograph
Change in non-invasive tear film break-up time from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Non-invasive tear film break-up time will be evaluated using Keratograph
Change in light dispersion from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Light dispersion will be evaluated using the Optical Quality Analysis System
Change in cytokine levels from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Cytokine leves will be evaluated using immunoassay
Change in therapeutic compliance from baseline to 6 months after treatment | From baseline to 6 months after treatment
  Therapeutic compliance will be evaluated using Medication adherence rating scale (MARS). The total score ranges from 0-10 with a higher score indicating better adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burgos Blasco, MD, PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No